CLINICAL TRIAL: NCT07067320
Title: Efficacy of Bibliotherapy Combined With Games to Reduce Fear of the Dark in Young Children: Results From a Clinical Trial
Brief Title: Bibliotherapy Combined With Games to Reduce Fear of the Dark in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Mireia Orgilés Amorós, Dr., Universidad Miguel Hernandez de Elche
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DPS.MOA.210423
Record Dates: First submitted 2025-06-11; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Bibliotherapy; Fear of the Dark; Nighttime Fears
Keywords: Nighttime fears; Bibliotherapy; Psychological treatment; Clinical trial
MeSH Terms: conditions — Nyctophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group receiving bibliotherapeutic intervention (Experimental): Bibliotherapy combined with games to overcome fear of the dark
  Interventions: Behavioral: Bibliotherapy combined with games to overcome fear of the dark
- Waiting list control group (receiving intervention at the end of treatment with experimental group) (No Intervention)

INTERVENTIONS:
Behavioral: Bibliotherapy combined with games to overcome fear of the dark — Bibliotherapy combined with games, applied by parents at home. Treatment based on cognitive-behavioural techniques. Duration: 4-5 weeks. Experimental group recived this bibliotherapeutic intervention.
  Arms: Experimental group receiving bibliotherapeutic intervention

SUMMARY:
Intense fear of the dark is a common issue among children, which can interfere with their daily functioning at family, social, and academic levels. This study aims to analyse the effectiveness of a psychotherapeutic intervention based on bibliotherapy combined with play to overcome the fear of the dark in children between 4 and 8 years old. A total of 38 children participated, who were assigned to the experimental and control conditions on the waiting list. The bibliotherapy intervention in the experimental condition involved reading a book and playing the games proposed in each chapter. The intervention was applied by parents at home with their children (during 4-5 weeks) and contained cognitive-behavioural techniques, such as gradual in vivo exposure, relaxation techniques, modelling and positive reinforcement, among others. It is expected that children's nighttime fears will decrease significantly and there will be significant improvements in nighttime behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Being between 4 and 8 years old
* Obtaining a score of 32 or higher on the Parent Version of the Nighttime Fears Scale (NFS-P; Orgilés et al., 2024)

Exclusion Criteria:

* Not being within the established age range
* Scoring less than 31on the Parent Version of the Nighttime Fears Scale (NFS-P; Orgilés et al., 2024)

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Nighttime fears | Pre- and post-intervention assessment (treatment lasts 4-5 weeks). There will also be a follow-up assessment 12 months after the end of the intervention.
  Parent Version of the Nighttime Fears Scale (NFS-P): The NFS-P assesses school-age children's level of fear at night, as reported by their parents. It contains four subscales: fear of nighttime features and distressing experiences (stimuli associated with darkness), fear of loss or separation from family (loss or non-presence of attachment figures and other family members), fear of imaginary stimuli (non-factual stimuli that may be likely to cause fear) and fear of real stimuli. It consists of 21 items that ask about night-time situations that are likely to cause fear in children. These items have a 5-point response scale, ranging from 0 (Not at all) to 4 (Very much). The higher the score, the greater the intensity of night-time fears.

SECONDARY OUTCOMES:
Nighttime functioning | From enrollment to the end of treatment at 4-5 weeks
  On a daily basis, families completed a log on different behaviours of their children during the night. Variables included: number of minutes it takes to go to bed, number of minutes it takes to fall asleep, avoidance behaviours, need for company to fall asleep, presence of security light, number of night-time calls to parents' bed, number of night-time visits to parents' bed, whether they sleep in their bed all night and, finally, whether they made use of the book and/or games.
Nighttime functioning | Pre- and post-intervention assessment (treatment lasts 4-5 weeks). There will also be a follow-up assessment 12 months after the end of the intervention.
  Nighttime Behaviors Questionnaire for Children - Parent-reported (NBQC-P): The NBQC-P assesses, through parents' responses, children's usual behaviours before going to sleep and during the night. It consists of three subscales: need for company, problems during the night and problems going to sleep. It contains 13 items, with a Likert-type response scale from 0 (Never or almost never) to 4 (Always or almost always). A higher score on each dimension implies a greater need for company to sleep, greater resistance before going to bed and greater interference with night-time awakenings.
Adaptive nocturnal behaviours | Pre- and post-intervention assessment (treatment lasts 4-5 weeks). There will also be a follow-up assessment 12 months after the end of the intervention.
  What I Can Do At Night - Parent Form (WICDAN-P): It assesses, through parents, children's ability to perform adaptive night-time behaviours during the last week. The scale consists of 11 items, with a 3-point response scale (0 = No; 1 = Yes, with difficulty or hesitation; 2 = Yes, with ease). The total score of the questionnaire is from 0 to 22. A higher score indicates adaptive night-time behaviour.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Miguel Hernández, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the small sample size and the sensitive nature of children's psychological data, with the primary aim of ensuring confidentiality and anonymity.